CLINICAL TRIAL: NCT07145476
Title: Efficacy and Neurophysiological Correlates of a Bilateral Robotic Treatment for Patients With Chronic Stroke Outcomes
Brief Title: Bilateral Robotic Rehabilitation in Chronic Stroke
Acronym: BILAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmelo Chisari (Other)
Responsible Party: Sponsor-Investigator, Carmelo Chisari, Prof., Azienda Ospedaliero, Universitaria Pisana
Organization: Azienda Ospedaliero, Universitaria Pisana (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17605
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Robotic; Neuroplasticity; Personalized Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RHS (Experimental): Right Hemisphere affected
  Interventions: Device: Robotic arm exoskeleton integrated with cognitively engaging serious games
- LHS (Experimental): Left Hemisphere affected
  Interventions: Device: Robotic arm exoskeleton integrated with cognitively engaging serious games

INTERVENTIONS:
Device: Robotic arm exoskeleton integrated with cognitively engaging serious games — A specific sequence of exercises including passive and active- assisted movements, unilateral and bilateral reaching tasks with visual feedback and bimanual symmetric and asymmetric coordination tasks.

SUMMARY:
This study investigated the effectiveness and neurophysiological correlates of Bilateral Robot-Assisted Training (BRAT) in right-handed individuals with chronic unilateral stroke, focusing on how lesion side (dominant vs. non-dominant hemisphere) influences recovery. Twenty-four participants (>6 months post-stroke) completed a three-week BRAT program using the ALEx-RS robotic exoskeleton integrated with cognitively engaging serious games involving symmetric and asymmetric upper limb tasks.

Clinical outcomes (Fugl-Meyer Assessment, Bimanual Activity Test, Motricity Index) and kinematic measures (movement smoothness, movement duration) were assessed at baseline, post-treatment, and at two-month follow-up. Significant improvements (p < 0.05) in all outcomes were observed after training and maintained at follow-up.

Patients with left hemiparesis (non-dominant side affected) showed greater gains in movement smoothness and bimanual task quality, suggesting recovery of more physiological motor patterns. Conversely, those with right hemiparesis (dominant side affected) improved mainly in movement speed, indicating compensatory strategy use. Greater baseline impairment predicted larger kinematic gains, particularly in the left hemiparesis group.

These findings support BRAT as an effective intervention for chronic stroke and underscore the importance of lesion side in shaping recovery profiles, with implications for personalized rehabilitation planning.

ELIGIBILITY:
Inclusion Criteria:

* first-ever unilateral stroke event;
* upper limb paresis with the ability to perform at least antigravity movements of the upper limb;
* right- hand dominance.

Exclusion Criteria:

* impossibility to provide informed consent;
* cognitive impairment limiting the ability to understand the therapist's directions (screening Mini-Mental State Examination score <24/30);
* hemispatial neglect, severe memory/attention impairment or severe aphasia;
* degree of spasticity of the upper limb such as to make the use of robotic devices impossible (Modified Ashworth Scale score > 3).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Enrollment: 24 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Changes in Fugl-Meyer for the Upper Limb (UEFM) scale pre vs post training | From the pre-training evaluation (T0) to the post-training evaluation (T1), about 3 weeks after T0, to the follow up T2, about 2 months after T1
  The Fugl-Meyer for the Upper Limb ranges from 0 to 66, with higher scores indicating better performance
Changes in Motricity Index (MI) scale pre vs post training | From the pre-training evaluation (T0) to the post-training evaluation (T1), about 3 weeks after T0, to the follow up T2, about 2 months after T1
  The Motricity Index ranges from 0 to 100, with higher scores indicating better performance
Changes in Bimanual Activity Test (BAT) scale pre vs post training | From the pre-training evaluation (T0) to the post-training evaluation (T1), about 3 weeks after T0, to the follow up T2, about 2 months after T1
  The Bimanual Activity Test ranges from 0 to 100, with higher scores indicating better performance

SECONDARY OUTCOMES:
Changes in movement smoothness pre vs post training | From the pre-training evaluation (T0) to the post-training evaluation (T1), about 3 weeks after T0
  The smoothness of patients' movements during reaching tasks with the exoskeleton will be measured using the modified Spectral ARC length (SPARC), with higher scores indicating better performance
Changes in movement duration pre vs post training | From the pre-training evaluation (T0) to the post-training evaluation (T1), about 3 weeks after T0
  The duration of patients' movements during reaching tasks with the exoskeleton will be measured in seconds, with shorter durations indicating better performance

CONTACTS AND LOCATIONS:
Locations (1):
- AOUP, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No